CLINICAL TRIAL: NCT01216189
Title: Sexual Function and Wellbeing in Females Diagnosed With Rectal Cancer
Brief Title: Sexual Function and Wellbeing in Females With Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Swedish Cancer Society (Other)
Responsible Party: Principal Investigator, Anna Martling, Professor, Senior Consultant Surgeon, Karolinska Institutet
Other Study IDs: 2008/247-31/3
Record Dates: First submitted 2010-10-04; First posted 2010-10-07 (Estimated); Results first posted 2021-04-09 (Actual); Last update posted 2021-04-09 (Actual); Status verified 2021-04

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Preoperative radiotherapy; Pelvic surgery; Sexual function; Wellbeing; Hormone levels
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Preoperative radiotherapy: Women with rectal cancer treated with preoperative radiotherapy (RT) and surgery.
  Interventions: Radiation: Preoperative radiotherapy
- No preoperative radiotherapy: Women with rectal cancer treated with surgery alone (no RT).

INTERVENTIONS:
Radiation: Preoperative radiotherapy — Preoperative radiotherapy (RT) was administered as either short course (5Gy x5) or long-course (2Gy x25 or 1.8 Gy x25 with or without 3 fractions of boost to the primary tumor and radiologically malignant lymph nodes) treatment with or without concomitant or sequential chemotherapy. Oncological treatment was decided at a multidisciplinary team conference.
  Groups: Preoperative radiotherapy

SUMMARY:
Preoperative radiotherapy (RT) and pelvic surgery is recommended to many patients with rectal cancer. For women there are theoretical reasons to believe that the treatment may affect hormone levels, sexual function and wellbeing. To address these questions a longitudinal observational study was initiated where androgen levels and sexual function were assessed before treatment (baseline) and during a follow-up period of two years.

DETAILED DESCRIPTION:
Women with rectal cancer stage I to III planned for abdominal surgery was included in the study. Women treated with preoperative RT were assigned to the exposed group and women treated with surgery alone were assigned to the unexposed group.

142 participants were enrolled at five outpatient rectal cancer centres in Sweden between 2008 and 2013. Patient data, fasting venous blood samples and questionnaires regarding sexual function and well-being were collected at a baseline visit before start of oncologic treatment, 1 year after surgery and 2 years after surgery (only questionnaires). Women treated with preoperative RT for rectal cancer had an additional venous blood sample taken the day before surgery.

Changes in serum levels of testosterone and sexual function during follow-up was assessed and compared between exposed and unexposed participants.

ELIGIBILITY:
Inclusion Criteria:

* Females diagnosed with rectal cancer stadium I-III, planned surgery with or without preoperative radiotherapy.

Exclusion Criteria:

* Rectal cancer stadium IV
* Previous radiotherapy to the pelvic region
* Inability to provide informed consent.
* Life expectancy less than 2 years.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Females with rectal cancer stadium I-III, planned for abdominal surgery, with or without preoperative radiotherapy.
Sampling Method: Probability Sample
Enrollment: 142 (Actual)
Dates: Start 2008-06; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Martling, Principal Investigator — Karolinska Institutet
Locations (5):
- Sweden (5):
  - Linköping University Hospital, Linköping
  - Norrköping Hospital, Norrköping
  - Örebro University Hospital, Örebro
  - Ersta Hospital, Stockholm
  - Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segelman J, Martling A, Machado M, Holm T, Bergmark K, Floter Radestad A. Preoperative sexual function in women with rectal cancer. Eur J Surg Oncol. 2013 Oct;39(10):1079-86. doi: 10.1016/j.ejso.2013.07.091. Epub 2013 Aug 15. PMID 23953232
- [Result] Segelman J, Buchli C, Svanstrom Rojvall A, Matthiessen P, Arver S, Bottai M, Ahlberg M, Jasuja R, Floter-Radestad A, Martling A. Effect of radiotherapy for rectal cancer on ovarian androgen production. Br J Surg. 2019 Feb;106(3):267-275. doi: 10.1002/bjs.10980. Epub 2018 Sep 12. PMID 30277569
- [Result] Svanstrom Rojvall A, Buchli C, Bottai M, Ahlberg M, Floter-Radestad A, Martling A, Segelman J. Effect of radiotherapy for rectal cancer on female sexual function: a prospective cohort study. Br J Surg. 2020 Apr;107(5):525-536. doi: 10.1002/bjs.11373. Epub 2019 Dec 3. PMID 31792944

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from five Swedish outpatient rectal cancer centres in Sweden (Karolinska University Hospital, Ersta Hospital, Örebro University Hospital, Linköping University Hospital and Norrköping Hospital) between June 2008 and August 2013. Of 404 women with rectal cancer assessed for eligibility, 142 were included in the study.
Period: Overall Study
Arm/Group | Preoperative Radiotherapy | No Preoperative Radiotherapy
Started | 110 | 32
Completed | 85 | 27
Not Completed | 25 | 5
Not completed — Lost to Follow-up | 21 | 3
Not completed — Death | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preoperative Radiotherapy | No Preoperative Radiotherapy | Total
Number analyzed (Participants) | 110 | 32 | 142
Age, Continuous [Median (Full Range); unit: years] | 62 [26 to 81] | 69 [46 to 90] | 65.5 [26 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 32 | 142
  Male | 0 | 0 | 0
BMI [Median (Full Range); unit: kg/m2] | 24.2 [17.3 to 37.4] | 24.4 [18.2 to 39.5] | 24.3 [17.3 to 39.5]
ASA score [Count of Participants; unit: Participants] — ASA score is a classification system for physical status ranging from scores I to VI with higher scores indicating worse physical status. Definitions of scores: I = Normal healthy person, II = A patient with mild systemic disease, III = A patient with severe systemic disease.
  Participants
    I | 35 | 7 | 42
    II | 58 | 13 | 71
    III | 16 | 9 | 25
    Missing | 1 | 3 | 4
Tumour distance from anal verge [Count of Participants; unit: Participants]
  0-4 cm | 45 | 4 | 49
  5-10 cm | 40 | 14 | 54
  11-15 cm | 23 | 12 | 35
  Missing | 2 | 2 | 4
Type of preoperative RT [Count of Participants; unit: Participants]
  Short course (5Gy x5) | 73 | 0 | 73
  Long course (2 Gy x25 or 1.8 x28) | 37 | 0 | 37
  No RT | 0 | 32 | 32
Type of Surgery [Count of Participants; unit: Participants]
  Anterior resection | 54 | 20 | 74
  Abdominal excision | 53 | 8 | 61
  No abdominal surgery | 2 | 2 | 4
  Missing | 1 | 2 | 3
Resection of gynaecological organs [Count of Participants; unit: Participants] — Includes resections before study inclusion and as part of rectal cancer surgery.
  Participants
    Hysterectomy | 13 | 5 | 18
    Unilateral/bilateral oophorectomy | 16 | 4 | 20
    Partial vaginal resection | 9 | 0 | 9
    No resection | 71 | 21 | 92
    Missing | 1 | 2 | 3
Pathological tumour stage [Count of Participants; unit: Participants] — Pathological tumour stage is determined by examining tissue removed during surgery. Staging is based on the American Joint Committee on Cancer (AJCC) TNM system, with T being the extent of the tumour, N spread to nearby lymph nodes and M spread to distant sites. This is summarised into a score ranging from 0 to IV, with 0 being very early cancer and higher numbers indicating more advanced cancer.
  Participants
    0 | 10 | 1 | 11
    I | 24 | 8 | 32
    II | 29 | 6 | 35
    III | 39 | 13 | 52
    IV | 4 | 1 | 5
    Missing | 4 | 3 | 7
Neoadjuvant chemotherapy [Count of Participants; unit: Participants]
  Yes | 35 | 1 | 36
  No | 74 | 29 | 103
  Missing | 1 | 2 | 3
Adjuvant chemotherapy [Count of Participants; unit: Participants]
  Yes | 36 | 9 | 45
  No | 73 | 21 | 94
  Missing | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Serum Testosterone Levels Between Baseline and 1 Year After Surgery.
Description: Fasting venous blood samples were collected at baseline visit (prior to oncological treatment) and 1 year follow-up. Participants treated with preoperative radiotherapy (RT) had an additional blood sample taken the day before surgery. Serum testosterone levels (T) were measured with liquid chromatography-mass spectrometry using the LC-MS/MS Quattro Premier Xevo TQ MS (Waters Corporation, Milford, MA, USA). The total coefficients of variation (CVtot) were 7% at 2.8 nmol/L and 6% at 15 nmol/L.
Time Frame: Baseline, the week before surgery and 1 year after surgery.
Population: 17 of the included 142 participants were excluded due to history of oophorectomy, resulting in 125 participants analysed. Participants in the group "No preoperative radiotherapy" had no blood samples taken at the time point "After RT/before surgery".
Measure: Median (Full Range); unit: nmol/l
Arm/Group | Preoperative Radiotherapy | No Preoperative Radiotherapy
Number analyzed (Participants) | 98 | 27
nmol/l
  Baseline | 0.6 [0.1 to 3.6] | 0.6 [0.2 to 4.8]
  After RT/before surgery: number analyzed (Participants) | 87 | 0
  After RT/before surgery | 0.6 [0.2 to 3.8] |
  1 year after surgery: number analyzed (Participants) | 66 | 20
  1 year after surgery | 0.5 [0.1 to 2.3] | 0.6 [0.2 to 1.3]
Statistical Analysis 1: Comparison: Preoperative Radiotherapy; The change in serum testosterone levels between baseline and 1 year was assessed using longitudinal regression analysis (GEE); Test type: Superiority; p = 0.004, Regression, Linear — The threshold for statistical significance was p = 0.05; Model adjusted for menopausal status; Mean change = -0.138, 95% CI 2-sided [-0.232 to -0.044]
Statistical Analysis 2: Comparison: No Preoperative Radiotherapy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.805, Regression, Linear — The threshold for statistical significance was p=0.05; Model adjusted for menopausal status; Mean change = -0.011, 95% CI 2-sided [-0.097 to 0.075]

2. Primary Outcome: Change in Sexual Function (Total FSFI Scores) Between Baseline and 2 Years Follow-up.
Description: Sexual function was assessed using the Female Sexual Function Index (FSFI). The FSFI questionnaire is a 19-item multiple-choice, self-assessment tool validated for use in the general population as well as for patients with cancer. It covers six domains of sexual function in women; desire (2 items), arousal (4 items), lubrication (4 items), orgasm (3 items), satisfaction (3 items) and pain (3 items). Items scores between 0 or 1 to 5, with lower scores indicating worse function. A total FSFI score can be calculated when all items are completed. Minimal total score is 4 points and maximal score is 95 points, with lower scores indicating worse function. A total FSFI score of less than 26.55 points was used to define overall sexual dysfunction.
Time Frame: Baseline, 1 year after surgery and 2 years after surgery.
Population: Of the 142 participants included in the study, 3 were excluded due to not answering FSFI questionnaires at any timepoint. Total FSFI scores were only calculated for available questionnaires without missing items.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Preoperative Radiotherapy | No Preoperative Radiotherapy
Number analyzed (Participants) | 109 | 30
score on a scale
  Baseline: number analyzed (Participants) | 89 | 25
  Baseline | 18.5 [2.0 to 36.0] | 6.7 [2.0 to 30.7]
  1 year after surgery: number analyzed (Participants) | 79 | 21
  1 year after surgery | 11.1 [2.0 to 34.5] | 5.8 [2.0 to 33.3]
  2 years after surgery: number analyzed (Participants) | 53 | 12
  2 years after surgery | 10.8 [2.0 to 34.8] | 6.5 [2.3 to 31.7]
Statistical Analysis 1: Comparison: Preoperative Radiotherapy vs No Preoperative Radiotherapy; The association between mean change in total FSFI score and preoperative RT was assessed using longitudinal regression analysis (GEE), using "no preoperative radiotherapy" as the reference group; Test type: Superiority; p = 0.013, Regression, Linear — The threshold for statistical significance was p=0.05; Model adjusted for Age, Psychological General Well-being total score and relationship with partner; Mean change in FSFI scores = -9.33, 95% CI 2-sided [-16.66 to -1.99]

ADVERSE EVENTS:
Description: Adverse Events were not monitored.
Groups:
- Preoperative RT: Women with rectal cancer treated with preoperative radiotherapy (RT) and surgery.
- No Preoperative RT: Women with rectal cancer treated with surgery alone (no RT).
Arm/Group | Preoperative RT | No Preoperative RT
All-Cause Mortality (participants affected / at risk) | 4/110 | 2/32
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes